CLINICAL TRIAL: NCT07236606
Title: A Phase 3, Open-Label Study to Evaluate the Efficacy, Safety, and Pharmacodynamics of RGX 121 in Pediatric Participants With Neuronopathic MPS II (Hunter Syndrome)
Brief Title: RGX-121-3102 Gene Therapy in Participants With MPS II (Hunter Syndrome)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGX-121-3102
Record Dates: First submitted 2025-11-05; First posted 2025-11-19 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: MPS II; Hunter Syndrome (MPS II)
Keywords: Mucopolysaccharidosis II; Gene Therapy
MeSH Terms: conditions — Sudden Infant Death; Mucopolysaccharidosis II

STUDY DESIGN:
Intervention Model Description: Dose Escalation
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 2.9×1011 GC/g brain mass of RGX 121 (Experimental): AAV9.CB7.hIDS
  Interventions: Genetic: RGX-121-3102

INTERVENTIONS:
Genetic: RGX-121-3102 — Recombinant adeno-associated virus serotype 9 [AAV9] capsid containing human iduronate-2-sulfatase (hIDS) expression cassette

SUMMARY:
RGX-121 is a gene therapy which is intended to deliver a functional copy of the iduronate-2-sulfatase gene (IDS) to the central nervous system. This study is a safety, efficacy, and pharmacodynamic dose ranging study to determine whether RGX-121 is safe, effective and well-tolerated by patients with MPS II (Hunter Syndrome)

DETAILED DESCRIPTION:
MPS II (Hunter Syndrome) is a rare X-linked recessive genetic disease caused by mutations in the iduronate-2-sulfatase gene (IDS). Enzyme replacement therapy (ERT) with recombinant idursulfase (ELAPRASE®) is the only approved product for the treatment of Hunter syndrome; however, ERT as currently administered does not cross the blood brain barrier and is therefore unable to address the unmet need in MPS II patients with central nervous system (CNS) (neurodevelopment and behavior) involvement. RGX-121 is designed to deliver a functional gene to cells in the CNS. Iduronate-2-sulfatase (I2S) may then be secreted by transduced cells, which may then cross-correct non-transduced cells by taking up the functional enzyme. This is a Phase III, open-label, confirmatory study investigating the efficacy, safety, and pharmacodynamics of RGX-121 treatment of patients with neuronopathic mucopolysaccharidosis type II (MPS II) aged ≥ 4 months to less than 5 years. A one time dose of RGX-121 will be studied in 2 male pediatric participants with neuronopathic MPS II, as supplemented in the analysis with 13 participants who were separately analyzed in the pivotal RGX-121-101 Part 2 study.

ELIGIBILITY:
Inclusion Criteria:

* The participant's legal guardian(s) is (are) willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any study-related procedures being performed.
* Is a male ≥ 4 months to < 5 years of age on Day 1.
* Has a documented diagnosis of MPS II, with a confirmed neuronopathic phenotype.
* Has a BSID-III Cognitive Composite score at or below -1SD (85) from the normative mean.
* Has 2 consecutive neurodevelopment assessments that support a decline on MSEL Visual Reception, Expressive Language, or Fine Motor, or BSID-III Cognitive, Expressive Communication, or Fine Motor of ≥ 1 SD on serial neurodevelopment testing administered between 3 to 36 months apart. Evidence for neurodevelopmental decline can be provided from historical medical records.
* Has a relative clinically diagnosed with neuronopathic MPS II who has the same IDS variant(s) as the participant AND the participant, in the opinion of a geneticist, has inherited a neuronopathic form of MPS II. Evidence for support of a relative with neuronopathic MPS II should be provided through medical record documentation of neurodevelopmental function at or below -2 SD from the normative mean. If standard scores are unavailable to document SD from the normative mean, a developmental quotient (AEq/chronological age × 100) of ≤ 60 can be used to document neuronopathic MPS II.
* Has documented variant(s) in IDS known to result in a neuronopathic phenotype. The participant's neuronopathic phenotype will be confirmed by an independent genetic review, with documented supporting evidence from previously reported cases of the same variant(s).
* Has sufficient auditory and visual capacity, with or without aids, to complete the required protocol testing, and be compliant with wearing the aid, if applicable, on testing days.
* Able to ambulate 100 meters independently without use of assistive devices, if the participant is, based on the judgement of the investigator, of a chronological age at screening at which independent ambulation would typically be expected in a child with neuronopathic MPS II.
* Provision of signed and dated informed consent form (ICF) and willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* Has a contraindication for an intracisternal (IC) and intraventricular (IVR) infusion, including any of the following:
* Review of baseline MRI testing by the team of neuroradiologist/neurosurgeons participating in study shows a contradiction for an IC and IVR infusion.
* History of prior head/neck surgery, which resulted in a contraindication to both IC and IVR infusion, based on review of available information by the team of neuroradiologists/neurosurgeons participating in the study.
* Has any contradiction to computed tomography or general anesthesia.
* Has any contradiction to MRI or gadolinium.
* Has renal insufficiency as determined by an estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2, based on creatinine. If the laboratory determines that creatinine is less than the lower limit of assay validation or detection, then the lowest limit cutoff value will be used to estimate eGFR.
* Has previously experienced a clinically significant intracranial bleed that, in the opinion of the investigator and team of neuroradiologists/neurosurgeons, is a contraindication to IC and IVR infusion.
* Has an elevated intracranial pressure (≥ 30 cm H2O).
* Has any neurocognitive deficit not attributable to MPS II or diagnosis of a neuropsychiatric condition that may, in the opinion of the investigator, confound interpretation of study results.
* Has any contraindication to lumbar puncture.
* Has a (cerebral) ventricular shunt that in the opinion of the site neuroradiologist/ neurosurgeon and through discussion with the Medical Monitor, may impact the administration and proper dosing of the participant.
* Has had prior treatment with AAV-based gene therapy product.
* Has undergone HSCT.
* Is receiving idursulfase (ELAPRASE) via IT administration, or a blood brain barrier-crossing ERT. Participants receiving IT ELAPRASE or a blood brain barrier-crossing ERT may enroll if they agree to discontinue these therapies starting at least 3 months prior to dosing with RGX-121, and for the duration of follow-up.
* Has received idursulfase (ELAPRASE) IV and experienced a serious hypersensitivity reaction, including anaphylaxis, deemed related to IV idursulfase (ELAPRASE) administration. If the participant has experienced a severe hypersensitivity reaction, they may enroll in the trial if the hypersensitivity has been treated and the investigator, Medical Monitor, and Sponsor agree that it no longer poses a safety or efficacy risk.
* Has received any Investigational Product within 30 days of Day 1 or 5 half-lives before signing of the ICF, whichever is longer.
* Has any history of lymphoma or history of another cancer, other than squamous cell or basal cell carcinoma of the skin, that has not been in full remission for at least 1 year before Screening.
* Has a history of human immunodeficiency virus (HIV) or hepatitis B or hepatitis C virus (HCV) infection, or positive screening tests for hepatitis B surface antigen or hepatitis B core antibody, or hepatitis C (either hepatitis C antibody or HCV RNA) or HIV antibodies.
* Has a clinically significant ECG abnormality that, in the opinion of the investigator, would compromise the participant's safety.
* Has a serious or unstable medical or psychological condition that, in the opinion of the investigator, would compromise the participant's safety or successful participation in the study or interpretation of study results.
* Has uncontrolled seizures that in opinion of the investigator would put the participant at undue risk.
* Has uncontrolled hypertension despite medical treatment, defined for children ≤ 17 years of age to be systolic blood pressure (SBP) or diastolic blood pressure (DBP) > 99th percentile plus 5mmHg based on normative standards for age, sex, and height.
* Has a platelet count < 100,000 per µL.
* Has ALT or AST > 3 × ULN or total bilirubin > 1.5 × ULN at Screening unless the participant has a previously known history of Gilbert's syndrome.
* Is a first-degree family member of a clinical site employee or of any other individual involved with the conduct of the study.
* REGENXBIO staff involved in the planning and/or conduct of the study.
* Employees of the study site or any other individuals involved with the conduct of the study or immediate family members of such individuals.
* Has any condition that would contraindicate treatment with methylprednisolone, prednisone, tacrolimus, or sirolimus.
* Has a history of a hypersensitivity reaction to methylprednisolone, tacrolimus, sirolimus, or prednisone.
* Has a history of a primary immunodeficiency (eg, common variable immunodeficiency syndrome), splenectomy, or any underlying condition that predisposes the participant to infection.
* Has herpes zoster (varicella zoster virus [VZV]), CMV, or EBV infection that has not completely resolved at least 12 weeks prior to Screening.
* Has any infection requiring hospitalization or treatment with parenteral anti-infectives not resolved at least 8 weeks prior to Day -2.
* Has any active infection requiring oral anti-infectives (including antivirals) within 10 days prior to Day -2.
* Has a history of active tuberculosis (TB) or a positive Quantiferon-TB Gold test during Screening.
* Has any live, replication-competent vaccine within 6 weeks prior to Day-2.
* Had major surgery within 8 weeks before signing the ICF or major surgery planned during the study period.
* Anticipates the need for adenoidectomy or tonsillectomy within 6 months of enrollment. If adenoidectomy or tonsillectomy is anticipated, it should be performed prior to Screening.
* Has an absolute neutrophil count (ANC) < 1.0 × 103/µL.
* Has any condition or laboratory abnormality that the investigator believes would not be appropriate for immunosuppressive therapy.

Ages: 4 Months to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male
Enrollment: 2 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2031-05-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of RGX-121 on Neurodevelopmental Function (as measured by the Bayley Scales of Infant and Toddler Development, 3rd Edition) | Month 24
  To evaluate the effect of RGX-121 on the neurodevelopmental function as measured by the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III).
Efficacy of RGX-121 on Neurodevelopmental Function (as measured by Kaufman Assessment Battery for Children, 2nd Edition) | Month 24
  To evaluate the effect of RGX-121 on the neurodevelopmental function as measured by the Kaufman Assessment for Children, 2nd edition (KABC-II). The KABC-II is only given if the participant achieved the max ceiling on the BSID-III Cognitive scale at two consecutive administrations.
Long-term Safety of RGX-121 | Year 5
  To evaluate the safety of RGX-121 for up to five years including serious and adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) (Version 5.0)

SECONDARY OUTCOMES:
RGX-121 Change in CSF Biomarkers (as measured by D2S6) | Week 16, Week 52, Month 24
  To assess the effect of RGX-121 on Glycosaminoglycan (GAG) levels in CSF as measured by D2S6.
RGX-121 Effect on Daily Living Skills | Month 24
  Change from baseline on daily living skills as measured by the Vineland Adaptive Behavior Scales, 2nd Edition (VABS-II), Comprehensive Interview Form. The Vineland Adaptive Behavior Scale II (VABS-II) is a standardized paediatric functional assessment tool. The VABS-II offers a way to measure personal and social self-sufficiency in real-life situations and to observe how these cognitive abilities impact the autonomy management process when put into practice. The VABS-II consists in a semi-structured interview with the parents. Higher scores mean a better outcome.
RGX-121 Change in Brain Volume | Week 52 and Month 24
  To evaluate the efficacy of RGX-121 on the participant's change in brain volume of gray and white matter.
RGX-121 Effect on Auditory Capacity | Month 24
  To assess the effect of RGX-121 on change in auditory capacity measured by ABR testing from baseline.
RGX-121 Change in Urine Biomarkers (GAGs) | Week 52 and Month 24
  To assess the effect of RGX-121 on ERT-naïve, ERT- continuing participants and ERT-withdrawn participants GAGs levels in urine.
RGX-121 Safety | Month 24
  To evaluate the safety of RGX-121 for up to two years including adverse event reporting, laboratory evaluations, vital signs, physical examinations, and neurological assessments.
RGX-121 Change in CSF Biomarkers (I2S) | Week 52 and Month 24
  To assess the effect of RGX-121 on I2S in cerebral spinal fluid (CSF)
RGX-121 Change in Plasma Biomarkers (GAGs) | Week 52 and Month 24
  To asses the effect of RGX-121 on GAGs levels in plasma.
RGX-121 Change in Plasma Biomarkers (I2S) | Week 52 and Month 24
  To assess the effect of RGX-121 on I2S levels in plasma.
RGX-121 Long-term Change in Neurodevelopmental Parameters | Year 5
  Change from baseline in neurodevelopment parameters of cognitive, behavioral and adaptive function as measured by the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III) or Kaufman Assessment Battery for Children, 2nd Edition (KABC-II).
RGX-121 Long-term Change in CSF Biomarkers (D2S6) | Year 5
  To assess the long-term effect of RGX-121 on GAG levels in CSF as measured by D2S6.
RGX-121 Long-term Change in CSF Biomarkers (I2S) | Year 5
  To assess the long-term effect of RGX-121 on I2S levels in CSF.
RGX-121 Long-term Change in Plasma Biomarkers (GAGs) | Year 5
  To assess the long-term effect of RGX-121 on GAGs levels in plasma.
RGX-121 Long-term Change in Plasma Biomarkers (I2S) | Year 5
  To assess the long-term effect of RGX-121 on I2S levels in Plasma.
RGX-121 Long-term Effect on Auditory Capacity | Year 5
  To assess the long-term effect of RGX-121 on change in auditory capacity measured by ABR testing from baseline to Year 5.
RGX-121 Long-term Effect on Urine Biomarkers | Year 5
  To assess the long-term effect of RGX-121 on ERT-naïve, ERT- continuing participants and ERT-withdrawn participants GAGs levels in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Schramm, Study Director — St. Peters University Hospital
Locations (1):
- St. Peter's University Hospital, New Brunswick, New Jersey, United States